CLINICAL TRIAL: NCT02125071
Title: An Exploratory Clinical Trial to Evaluate the Pharmacokinetic Characteristics of I.V. Hepabig Injection Used for Prevention of Hepatitis B Relapse After Liver Transplantation
Brief Title: Study on the Pharmacokinetic Characteristics of I.V. Hepabig Injection Used for Prevention of Hepatitis B Relapse After Liver Transplantation
Acronym: LT
Status: Completed | Type: Observational
Sponsor: Dong-Gu Kim (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Sponsor-Investigator, Dong-Gu Kim, MD, Phd, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: I.V. Hepabig injection_IIT
Record Dates: First submitted 2014-03-31; First posted 2014-04-29 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Liver Cirrhosis; Chronic Hepatitis B
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepabig: Those who receiving I.V. Hepabig injection used for prevention of hepatitis B relapse after liver transplantation
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Blood Sample Collection before and after the administration of I.V. Hepabig Inj. on LT day(0 day); 1 day after; 1, 4, 12 and 24 weeks after LT.

SUMMARY:
An exploratory clinical trial to evaluate the pharmacokinetic characteristics of I.V. Hepabig injection used for prevention of hepatitis B relapse after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≤18 years old
* Patients who understand the informed consent form and signed the form voluntarily
* Patients who underwent liver transplantation due to HBV related disease and will be treated for prevention of hepatitis B relapse after liver transplantation

Exclusion Criteria:

* Multi-organ recipient or reimplantation
* IgA Deficiency
* Serious nephropathy
* Serious cardiovascular system failure within 6 months
* Ischemic or hemolytic anemia
* Condition of immunosuppression and immunodeficiency
* Hypersensitivity or allergic to blood products
* HIV or HCV positive
* Participation to other clinical trial within 3 months
* Pregnancy or breast feeding
* Those who the investigator determines inappropriate to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who receiving I.V. Hepabig injection for prevention of hepatitis B relapse after liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
anti-HBs titer | up to 6 months
  The anti-HBs titer is measured on the day of LT, day 1, week 1, week 4, week 12 and week 24, to determine the pharmacokinetic characteristic of Hepabig I.V. injection

CONTACTS AND LOCATIONS:
Overall Officials: Dong Gu Kim, MD, PhD, Principal Investigator — The Catholic University, Seoul St Mary Hospital
Locations (1):
- The Catholic University, Seoul St Mary Hospital, Seoul, Seoul, South Korea